CLINICAL TRIAL: NCT06082947
Title: αβT Cell/CD19+ B Cell Depletion for Alternative Donor Allogeneic Hematopoietic Cell Transplantation (HSCT) for Children and Young Adults With Hematologic Malignancies
Brief Title: αβT Cell/CD19+ B Cell Depletion for Alternative Donor Allogeneic Hematopoietic Cell Transplantation (HSCT)
Acronym: TB19DHCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB19DHCT
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hematopoietic Stem Cell Transplantation; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- HSCT using TCR αβ/CD19+ depleted grafts (Experimental): Allogeneic HSCT using the TCR αβ/CD19+ depleted platform and grafts from alternative donors (MUD, MMUD and haploidentical)
  Interventions: Device: CliniMACS®

INTERVENTIONS:
Device: CliniMACS® — CliniMACS® αβT cell/CD19+B cell depletion device for Children and Young Adults with Hematologic Malignancies undergoing alternative Donor Allogeneic Hematopoietic Cell Transplantation (HSCT)

SUMMARY:
This is a study utilizing the Magnetic-activated cell sorting (CliniMACS®) Alpha-Beta T-cell (αβT)/Cluster of Differentiation 19 (CD19), also called B lymphocyte antigen CD19 depletion device for Children and Young Adults with Hematologic Malignancies undergoing alternative Donor Allogeneic Hematopoietic Cell Transplantation (HSCT). Patients will receive an allogenic HSCT from a matched unrelated donor (MUD), mismatch unrelated donor (MMUD) or a mismatched related (haploidentical) donor. Patients will receive a granulocyte-colony stimulating factor (G-CSF) ± Plerixafor donor mobilized peripheral stem cell donor transplant following CliniMACS® αβT cell/CD19+B cell depletion. Cluster of Differentiation 34 (CD34) and αβT cell content of the graft is determined based on the transplant indication.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 30 years
* Patients who will benefit from an allogenic stem cell transplant to treat underlying primary hematological malignancy and lacks a suitably available matched sibling donor.
* Karnofsky Index or Lansky Performance Scale ≥ 60 % on pre-transplant evaluation.
* Karnofsky scores must be used for patients > 16 years of age and Lansky scores for patients ≤ 16 years of age.
* Patient or legal guardian must give informed consent if patient is ≥ 18 years. Legal guardian must give informed consent (and patient must give assent if appropriate) if patient is < 18 years.
* Adequate organ function (within 4 weeks of initiation of preparative regimen). For patients receiving Myeloablative conditioning (MAC) on this platform, they should meet organ function to tolerate MAC. Similar if patients are receiving Reduced intensity conditioning (RIC).
* High resolution human leukocyte antigen (HLA) available

Exclusion Criteria:

* Patient does not have a suitable donor who is willing and able (meets donor criteria).
* Patient reports a history of allergic reactions to murine protein
* Pregnant or lactating females are ineligible as many of the medications used in this protocol could be harmful to unborn children and infants. Female patients of childbearing potential females ≥11 years of age or post- menarche and should have a negative pregnancy test
* Patients with HIV or uncontrolled fungal, bacterial or viral infections are excluded. Patients with history of fungal disease during induction therapy may proceed if they have a significant response to antifungal therapy with no or minimal evidence of disease remaining by CT evaluation. Viremia by Pluripotency Check (PCR) analysis is not considered an active infection but may require immediate viral prophylaxis. Patients with possible fungal infections must have had at least 2 weeks of appropriate anti-fungal therapy and be asymptomatic -
* Patients receiving umbilical cord blood and matched sibling donor transplants

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
One-year overall survival of patients undergoing allogeneic HSCT using the T-Cell Receptor (TCR) αβ/CD19+ depleted platform and grafts from alternative donors (MUD, MMUD and haploidentical) | 1 year
  One-year overall survival of patients undergoing allogeneic HSCT

SECONDARY OUTCOMES:
Neutrophil and platelet engraftment following TCR αβ/CD19+ depleted alternative donor (MUD, MMUD and haploidentical) HSCT | 100 days
  Neutrophil and platelet engraftment by day 100
Incidence of final status graft failure | 1 year
  Incidence of final status graft failure by 1 year
Incidence grade III-IV acute graft versus host disease (GVHD) | 1 year
  Incidence grade III-IV acute graft versus host disease (GVHD) by 1 year
Incidence of chronic GVHD | 1 year
  Incidence of chronic GVHD by 1 year
100 day and 1 year Transplant related mortality | 1 year
  100 day and 1 year Transplant related mortality by 1 year
1 year Event free survival | 1 year
  1 year Event free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States